CLINICAL TRIAL: NCT06044350
Title: A Phase II/III Study to Evaluate the Efficacy and Safety of BAT4406F Injection in Patients With Neuromyelitis Optica Lineage Disease
Brief Title: A Clinical Trial of BAT4406F Injection in Patients With Neuromyelitis Optica Spectrum Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAT-4406F-002-CR
Record Dates: First submitted 2023-07-31; First posted 2023-09-21 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Optic Neuromyelitis Spectrum Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group：BAT4406F (Experimental): RCP：Intravenous infusion; Dosage:500mg/time; Time of administration:The drug was given at D 1 and D 182 respectively OLP：Intravenous infusion; Dosage:500mg/time; Time of administration: After D1 dosing, Every 6 months to 1 times
  Interventions: Drug: BAT4406F Injection
- Control group：BAT4406F Placebos (Active Comparator): RCP：Intravenous infusion; Dosage:500mg/time; Time of administration:The drug was given at D 1 and D 182 respectively OLP：Intravenous infusion; Dosage:500mg/time; Time of administration: After D1 dosing, Every 6 months to 1 times
  Interventions: Drug: BAT4406F Placebos

INTERVENTIONS:
Drug: BAT4406F Injection — Intravenous infusion; Dosage:500mg/time
  Arms: Experimental group：BAT4406F
Drug: BAT4406F Placebos — Intravenous infusion; Dosage:500mg/time
  Arms: Control group：BAT4406F Placebos

SUMMARY:
This is a phase II/III multicenter, randomized, double-blind, placebo-controlled study, to investigate the efficacy and safety of BAT4406F injection in patients with neuromyelitis optica lineage disease (NMOSD) who are positive for aquaporin 4 antibody (AQP4-IgG) .

DETAILED DESCRIPTION:
This study was a phase II/III multicenter, randomized, double-blind, placebo-controlled study, which was divided into screening period (4 weeks) , randomized control period (RCP) , and open-label period (Olp)A total of 162 subjects were enrolled during the screening period and randomly assigned 2:1 to either the BAT4406F group or the placebo group after randomization on Day 1 of the RCP, subjects would receive BAT4406F (at a dose of 500mg) or placebo, intravenously, at D 1 and D 182, respectively.

If any of the following conditions occur, subjects can enter OLP from RCP: 1. Subjects who complete the 52-week RCP study without recurrence of NMOSD can enter Olp within 14 days after the end of the RCP study. 2. In the stage of RCP, NMOSD recurred. After rescue therapy, the patients with stable condition could enter OLP within 28 days after diagnosis. Subjects continued to participate in the RCP study if they were not identified by CEC as having a relapse upon examination. 3. When a protocol-defined first relapse event of 35 cases is observed, or when all 162 subjects have completed randomization and 12 months have elapsed since the first dose in the last of these subjects, or when recommended by the Independent Data Monitoring Committee (IDMC) , the RCP study should be stopped for enrolled subjects, and all enrolled subjects at the RCP stage should stop the RCP study within 14 days of entry into OLP, after which subjects will receive BAT4406F injection at the same dose as RCP, at d 1 of OLP. After termination of the RCP study with BAT4406F every 6 months, subjects were given the option of enrolling in the OLP study.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to the age of 18 and less than or equal to 65 patients, gender not limited;
2. Met the 2015 international NMO diagnostic panel (IPND) criteria for NMOSD, And AQP4-IGG positive patients
3. Screening before 2 times at least 2 years experience with clinical records of relapse，or experienced at least 1 clinically documented recurrence within 1 year prior to screening
4. For subjects who had a relapse before screening, symptoms needed to be stable for at least 4 weeks before randomization
5. Into the group of former dosage of corticosteroids under 30 mg and prednisone equivalent，and the trial drug must be used within a month after the withdrawal of hormones
6. The score of EDSS 7 or less
7. Has the fertility of men and women must agree during treatment and 6 months after the last dose of using effective birth control method;
8. Agreed to participate in trials, and books to sign the informed consent

Exclusion Criteria:

1. CD19 + b-cell count below the lower limit of normal, b-cell-scavenger drugs used 6 months before baseline or within 5 half-lives of the drug, whichever is older (including but not limited to Rituximab, enalizumab, etc.) ;
2. 6 months prior to the baseline used other monoclonal antibody therapy;Baseline used within five half-life before other biological preparation;
3. Used it for 3 months prior to the baseline McCaw phenol ester, azathioprine and methotrexate;6 months prior to the baseline using cyclophosphamide;Baseline before five half-life
4. Within a month before the filter used intravenous immunoglobulin (IVIG), plasma exchange (PE);
5. Within 4 weeks before screening received vaccine or live attenuated;Within 2 weeks before the baseline received inactivated vaccine;Baseline received within 4 weeks before the new coronavirus vaccine
6. In another clinical study and the baseline from the test drug treatment under three months or 5 half-life of the drug (the long time limit shall prevail);
7. This test for monoclonal antibody has a history of allergies, known in drug allergy patients;Serious drug allergy or for two or over two kinds of food or drugs；
8. 6 months prior to screening, except NMOSD need continuous oral or intravenous glucocorticoid dose > 20 mg/day of any more than 21 days
9. Abnormal liver, kidney and bone marrow reserve
10. HIV positive at HIV history or enrollment screening; History of hepatitis B Andor hepatitis C or Hepatitis B surface antigen (HBSAG) positivity at screening [ or Hepatitis B core antibody positive, hepatitis B surface antibody negative, Hepatitis B virus deoxynucleotides (HBV DNA) quantification exceeding normal range ] ; Or Hepatitis C virus (HCV) antibody positive [ with HCV-rna quantitation exceeding the normal range ] , Treponema pallidum antibody positive at the time of enrollment;
11. Comply with any of the following subjects a latent or active TB infection related standards:

    1. Current or past people with active TB;
    2. In history and/or physical examination during filter tip physical signs or symptoms of active TB;
    3. Recent close contact with people with active TB;
    4. At the time of screening, the positive result of TB infected T cells was found. A test could be repeated if the subject's first tb-infected t-cell test result was inconclusive, and the patient was excluded from this study if the test result was inconclusive (or positive) again.
12. Covid-19 infection was diagnosed with clinical symptoms or signs consistent with 2019 coronavirus (COVID-19) infection (eg, fever, dry cough, dyspnea, sore throat, and fatigue) within 4 weeks before screening or during screening, or upon appropriate laboratory testing (at the discretion of the investigator or in accordance with local regulations) . If COVID-19 infection is confirmed before screening, appropriate laboratory testing is required to confirm that the infection has been cured;
13. Suffering from metabolic, hematological, renal, hepatic, pulmonary, neuroendocrine, cardiac, infectious, gastrointestinal or other autoimmune diseases, the researchers believe there is an unacceptable risk to patients, or it may affect NMOSD assessment;
14. According to the researchers, there was a history of drug and alcohol abuse (drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 125 mL of wine) in the 12 months before screening；
15. Subjects who are unable to undergo an MRI scan (for example, are allergic to Gd-containing MRI contrast media, have a pacemaker, defibrillator, or other metallic object with internal or external limitations to performing an MRI scan) ;
16. Pregnant or lactating women, and screening or baseline pregnancy test positive female subjects;
17. Researchers think that the other does not fit to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics | RCP: Day7, Day14, Day28, Day56, Day84, Day112, Day140, Day182, Day280, Day364. OLP:D7, D28, Day84, Day182, Day280, Day364. Week 40+26n (n=1, 2, 3.....) , Week 52+26n (n=1, 2, 3.....). And OLP maximum period for 3 years
  The follow-up time point of peripheral blood before and after the analysis to the medicine CD19 + B lymphocytes proportion/count change
Pharmacodynamics | RCP:in Day84、Day182、Day280、Day364. OLP: in Day1、Day84、Day182、Day280、Day364 of every years.And OLP maximum period for 3 years
  Serum immunoglobulin (IgG and IgM) levels were measured.
Pharmacodynamics | RCP:in Day84、Day182、Day280、Day364. OLP: in Day1、Day84、Day182、Day280、Day364 of every years.And OLP maximum period for 3 years
  AQP4-IgG levels were measured.
Pharmacokinetics（PK） | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Cmax
Pharmacokinetics（PK） | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Tmax
Pharmacokinetics（PK） | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Cmin
Pharmacokinetics（PK） | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  AUC0-tau
Pharmacokinetics（PK） | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  t1/2
Pharmacokinetics（PK） | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  CL
Pharmacokinetics（PK） | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Vd
Immunogenicity evaluation | RCP:in Day84、Day181、Day252、Day364. OLP: in Day84、Day181、Day252、Day364 of every years.And OLP maximum period for 3 years
  Resistant antibody positive rate (ADA)
Immunogenicity evaluation | RCP:in Day84、Day181、Day252、Day364. OLP: in Day84、Day181、Day252、Day364 of every years.And OLP maximum period for 3 years
  The titers of Ada positive samples

SECONDARY OUTCOMES:
Vital signs | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Number of participants with abnormal vital signs
physical examination | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Number of participants with abnormal physical examination findings
Laboratory tests | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Number of participants with abnormal laboratory test results
electrocardiogram（ ECG ） | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Number of participants with abnormal ECG readings
Adverse events（AE） | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Adverse events (AE) is happening, is happening because of adverse events leading to withdrawal Adverse events associated with drugs The occurrence of Serious adverse events (SAE)
Injection site reactions | Through study completion,up to 49 months. And OLP maximum period for 3 years.
  Number of participants with injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjun Chen, Doctor, Principal Investigator — Huashan Hospital; Chunfeng Liu, Doctor, Principal Investigator — Second Affiliated Hospital of Suzhou University; Qun Xue, Doctor, Principal Investigator — First Affiliated Hospital of Suzhou University; Yan Jiang, Doctor, Principal Investigator — Anhui Provincial Hospital; Yuying Zhao, Doctor, Principal Investigator — Shandong University Qilu Hospital; Li Guo, Doctor, Principal Investigator — Second Hebei Medical University Hospital; Meini Zhang, Doctor, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University; Huan Yang, Doctor, Principal Investigator — The Central South University Xiang Ya Hospital; Daishi Tian, Doctor, Principal Investigator — Tongji hospital affiliated to Tongji Medical College; Yuming Xu, Doctor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Jianglong Tu, Doctor, Principal Investigator — Second Affiliated Hospital of Nanchang University; Wei Qiu, Doctor, Principal Investigator — The third hospital affiliated to sun yat-sen university; Yamei Tang, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Honghao Wang, Doctor, Principal Investigator — The First People's Hospital of Guangzhou; Xiaoling Luo, Doctor, Principal Investigator — Shenzhen city people's hospital; Aiyu Lin, Doctor, Principal Investigator — First Affiliated Hospital of Fujian Medical University; Chunming Xie, Doctor, Principal Investigator — China University Hospital of Southeast University; Xiang Li, Doctor, Principal Investigator — The first hospital affiliated to wenzhou medical college; Lan Tan, Doctor, Principal Investigator — Qingdao City Hospital; Fudong Shi, Doctor, Principal Investigator — Tianjin Medical University General Hospital; Juming Yu, Doctor, Principal Investigator — Afﬁliated Hospital of North Sichuan Medical College; Jun Guo, Doctor, Principal Investigator — The Second Affiliated Hospital of the PLA Air Force Military Medical University; Jiewen Zhang, Doctor, Principal Investigator — Henan Provincial People's Hospital; Yanghua Tian, Doctor, Principal Investigator — Second Affiliated Hospital of Anhui Medical University; Jing Ding, Doctor, Principal Investigator — Shanghai Zhongshan Hospital; Ping Chen, Doctor, Principal Investigator — Xianyang yanan university hospital co., LTD; Zunbo Li, Doctor, Principal Investigator — Xi'an high-tech Hospital Co. , Ltd.; Qihe Dai, Doctor, Principal Investigator — Jingzhou city central hospital; Dan Liu, Doctor, Principal Investigator — the first hospital of Baotou medicine college; Junyan Liu, Doctor, Principal Investigator — Hebei Medical University Third Hospital; Yiqi Wang, Doctor, Principal Investigator — Zhejiang Province People's Hospital; Bo Hu, Doctor, Principal Investigator — Xiehe hospital affiliated to tongji medical college; Yanbing Han, Doctor, Principal Investigator — First Affiliated Hospital of the Kunming Medical University; Feng Wang, Doctor, Principal Investigator — Wuxi city people's hospital; Zhanhua Liang, Doctor, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; Weihe Zhang, Doctor, Principal Investigator — Sino-Japanese Friendship Hospital; Xiangyang Zhu, Doctor, Principal Investigator — Nantong First People's Hospital; Xinfeng Liu, Doctor, Principal Investigator — The Chinese people's liberation army general hospital in eastern theater; Weidong Pan, Doctor, Principal Investigator — Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine; Wei Lu, Doctor, Principal Investigator — The Central South University Xiang YA II hospital; Huiyu Feng, Doctor, Principal Investigator — The first hospital affiliated to sun yat-sen university; Feng Gao, Doctor, Principal Investigator — The first hospital of Peking University; Yun Xu, Doctor, Principal Investigator — Drum tower hospital affiliated to nanjing university school of medicine
Locations (45):
- China (45):
  - The First Affiliated Hospital of the Baotou Medical College of Inner Mongolia University of Science and Technology, Baotou
  - Beijing Hospital, Beijing
  - China-japan friendship Hospital, Beijing
  - The first hospital of Peking University, Beijing
  - The Central South University Xiang Ya Hospital, Changsha
  - Xiangya 2nd hospital of central south university, Changsha
  - First affiliated hospital of chongqing medical university, Chongqing
  - The first affiliated hospital of Dalian Medical University, Dalian
  - First affiliated hospital of fujian medical university, Fuzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The first hospital affiliated to sun yat-sen university, Guangzhou
  - The first People's Hospital of Guangzhou, Guangzhou
  - The third hospital affiliated to sun yat-sen university, Guangzhou
  - People's Hospital of Zhejiang province, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Second Affiliated Hospital of Anhui Medical University, Hefei
  - Shandong University Qilu Hospital, Jinan
  - Jingzhou Central Hospital, Jingzhou
  - First Affiliated Hospital of the Kunming Medical University, Kunming
  - Second Affiliated Hospital of Nanchang University, Nanchang
  - Affiliated Hospital of North Sichuan Medical College, Nanchong
  - Drum Tower Hospital affiliated to Medical College of Nanjing University, Nanjing
  - Southeast university affiliated zhongda hospital, Nanjing
  - The Chinese people's liberation army general hospital in eastern theater, Nanjing
  - The first People's Hospital of Nantong, Nantong
  - Qingdao municipal hospital, Qingdao
  - Mount Hua Hospital affiliated to Fudan University, Shanghai
  - Shuguang hospital affiliated to Shanghai University of Traditional Chinese medicine, Shanghai
  - Zhongshan hospital affiliated to Fudan University, Shanghai
  - Shenzhen city people's hospital, Shenzhen
  - Second Hebei Medical University Hospital, Shijia Zhuang
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - First Affiliated Hospital of Suzhou University, Suzhou
  - The Second Affiliated Hospital of Suzhou University, Suzhou
  - The first hospital of shanxi medical university, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
  - The first hospital affiliated to wenzhou medical college, Wenzhou
  - Tongji hospital affiliated to tongji medical college huazhong university of science and technology, Wuhan
  - Xiehe hospital affiliated to tongji medical college huazhong university of science and technology, Wuhan
  - Wuxi city people's hospital, Wuxi
  - Second Affiliated Hospital of the People's Liberation Army Air Force Military Medical University, Xi'an
  - Xi'an high-tech Hospital Co. , Ltd., Xi'an
  - Yan 'an University Xianyang Hospital Co. , Ltd., Xianyang
  - Henan province people's hospital, Zhengzhou
  - Zhengzhou university first affiliated hospital, Zhenzhou